CLINICAL TRIAL: NCT01054807
Title: Non-Dispensing Evaluation of an Investigational Galyfilcon A Soft Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Collaborators: Coles-Brennan Pty Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-0915; CTN# 155/2009 (Registry Identifier: Therapeutics Goods Aministration (TGA))
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2017-06

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (6):
- GalyfilconHL/Galyfilcon8.7/Galyfilcon8.3 (Other): Galyfilcon A Habitual Lens (Active Comparator)/Galyfilcon A 8.7 BC (Experimental)/Galyfilcon A 8.3 BC (Experimental)
  Interventions: Device: Galyfilcon A Habitual Lens; Device: Galyfilcon A 8.7 BC (Investigational); Device: Galyfilcon A 8.3 BC (Investigational)
- Galyfilcon8.7/Galyfilcon8.3/GalyfilconHL (Other): Galyfilcon A 8.7 BC (Experimental)/Galyfilcon A 8.3 BC (Experimental)/Galyfilcon A Habitual Lens (Active Comparator)
  Interventions: Device: Galyfilcon A Habitual Lens; Device: Galyfilcon A 8.7 BC (Investigational); Device: Galyfilcon A 8.3 BC (Investigational)
- GalyfilconHL/Galyfilcon8.3/Galyfilcon8.7 (Other): Galyfilcon A Habitual Lens (Active Comparator)/Galyfilcon A 8.3 BC (Experimental)/Galyfilcon A 8.7 BC (Experimental)
  Interventions: Device: Galyfilcon A Habitual Lens; Device: Galyfilcon A 8.7 BC (Investigational); Device: Galyfilcon A 8.3 BC (Investigational)
- Galyfilcon 8.7/Galyfilcon HL/Galyfilcon 8.3 (Other): Galyfilcon A 8.7 BC (Experimental)/Galyfilcon A Habitual Lens (Active Comparator) /Galyfilcon A 8.3 BC (Experimental)
  Interventions: Device: Galyfilcon A Habitual Lens; Device: Galyfilcon A 8.7 BC (Investigational); Device: Galyfilcon A 8.3 BC (Investigational)
- Galyfilcon8.3/GalyfilconHL/Galyfilcon8.7 (Other): Galyfilcon A 8.3 BC (Experimental)/Galyfilcon A Habitual Lens (Active Comparator)/Galyfilcon A 8.7 BC (Experimental)
  Interventions: Device: Galyfilcon A Habitual Lens; Device: Galyfilcon A 8.7 BC (Investigational); Device: Galyfilcon A 8.3 BC (Investigational)
- Galyfilcon8.3/Galyfilcon8.7/GalyfilconHL (Other): Galyfilcon A 8.3 BC (Experimental)/Galyfilcon A 8.7 BC (Experimental)/Galyfilcon A Habitual Lens (Active Comparator)
  Interventions: Device: Galyfilcon A Habitual Lens; Device: Galyfilcon A 8.7 BC (Investigational); Device: Galyfilcon A 8.3 BC (Investigational)

INTERVENTIONS:
Device: Galyfilcon A Habitual Lens — Comparison of three soft contact lens designs.
Device: Galyfilcon A 8.7 BC (Investigational) — Comparison of three soft contact lens designs.
Device: Galyfilcon A 8.3 BC (Investigational) — Comparison of three soft contact lens designs

SUMMARY:
The purpose of this investigation is to compare the fit characteristics and vision attributes of an investigational Galyfilcon A contact lens and an approved Galyfilcon A contact lens.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age (i.e., at least 18 years old)
* Sign a written informed consent
* Have contact lens distance sphere requirement in the range -1.00D to -6.00D
* Have spectacle astigmatism <1.25D in each eye
* Currently wear ACUVUE® ADVANCE™ (for at least 6 months) with documentation of current prescription.
* Have normal eyes with no evidence of abnormality or disease.

Exclusion Criteria:

* Required concurrent ocular medication
* Any systemic illness which would contra-indicate lens wear or the medical treatment of which would affect vision or successful lens wear.
* Eye injury or surgery within eight weeks immediately prior to enrollment for this study.
* Abnormal lacrimal secretions
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Keratoconus or other corneal irregularity.
* Pregnancy, lactating or planning a pregnancy at the time of enrolment.
* Participation in any concurrent clinical trial
* Known allergy to silver, silver ions, or silver containing compounds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-11-01 (Actual); Primary Completion 2010-03-01 (Actual); Study Completion 2010-03-01 (Actual)

PRIMARY OUTCOMES:
Comparison of Lens Fit Characteristics | Approximately 40 minutes of wear time
  At the screening visit, the following baseline measurements will be taken of the subject's habitual contact lenses (Control):
  * Visual Acuity (logMar)
  * Over-refraction with Visual Acuity
  * Fit acceptability (acceptable/non-acceptable)
Evaluation of Inter-Changeability | Approximately 40 minutes of wear time
  In a bilateral fashion, the subject will wear Test/Control lens according to a pre-designed randomization schedule. Immediately upon insertion, the following variables will be assessed:
  * Ease of handling of the lenses- by Investigator
  * Comfort on insertion
  After 30-40 minutes of settling time the following variables will be collected:
  * Subjective comfort after settling
  * Visual Acuity (logMar)
  * Corneal coverage (Y/N)
  * Post-blink movement (mm)
  * Version Lag (mm)
  * Tightness on push-up (0-100 scale)
  * Overall fit acceptance (0-5 scale)
Determination of fit or Vision Differences | Approximately 40 minutes of wear time
  In a bilateral fashion, the subject will wear Test/Control lens according to a pre-designed randomization schedule. Immediately upon insertion, the following variables will be assessed:
  * Ease of handling of the lenses- by Investigator
  * Comfort on insertion
  After 30-40 minutes of settling time the following variables will be collected:
  * Subjective comfort after settling
  * Visual Acuity (logMar)
  * Corneal coverage (Y/N)
  * Post-blink movement (mm)
  * Version Lag (mm)
  * Tightness on push-up (0-100 scale)
  * Overall fit acceptance (0-5 scale)

CONTACTS AND LOCATIONS:
Overall Officials: Noel Brennan, McOptom PhD, Principal Investigator — Coles-Brennan Pty Ltd
Locations (1):
- Coles-Brennan Pty Ltd, Hawthorn, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No